CLINICAL TRIAL: NCT03870711
Title: 10% Lidocaine Spray for Pain Control During Intrauterine Device Insertion: A Randomized, Double-blinded, Placebo Controlled Trial
Brief Title: 10% Lidocaine Spray for Intrauterine Device Insertion
Acronym: LidocaineIUD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Si 240/2018
Record Dates: First submitted 2018-05-10; First posted 2019-03-12 (Actual); Last update posted 2020-01-30 (Actual); Status verified 2020-01

CONDITIONS: Contraception; Intrauterine Device
Keywords: Intrauterine device; lidocaine spray
MeSH Terms: interventions — Lidocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- group A (Experimental): 10% lidocaine spray
  Interventions: Drug: lidocaine spray
- group B (Placebo Comparator): sterile water
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: lidocaine spray — 10% lidocaine spray 4 puffs
  Other Names: Xylocaine
  Arms: group A
Drug: Placebo — Sterile water 4 puffs
  Other Names: Sterile water
  Arms: group B

SUMMARY:
Intrauterine device (IUD) insertion is a procedure that can cause pain. Fear of pain during IUD insertion is a barrier to use of this method. Currently, there is no recommended standard method for reducing pain during this procedure. From Cochrane Database 2015, some lidocaine formulations, such as lidocaine spray, lidocaine gel and lidocaine paracervical injection, could reduce pain during IUD insertion, but there is limited data on effect of lidocaine spray on reducing pain during insertion of IUD.

DETAILED DESCRIPTION:
Intrauterine device (IUD) is a high efficacy long-acting reversible contraceptive method. However, IUD insertion is a procedure that require well-trained medical personnel and can cause pain in several steps during insertion such as applying tenaculum, applying uterine sound and insertion of IUD. Fear of pain during IUD insertion is a barrier to use of this contraceptive method. Previous researches reported mean pain score with using visual analog scale (VAS) moderated pain (4.7/10 and 34.7-51.2/100). In several countries, pain control is used before IUD insertion procedure. Currently, there is no recommended standard method for reducing pain during this procedure. From Cochrane Database 2015, some lidocaine formulations, such as lidocaine spray, lidocaine gel and lidocaine paracervical injection, could reduce pain during IUD insertion, but there is limited data on effect of lidocaine spray on reducing pain during insertion of IUD.

Lidocaine is introduced to use for pain relieving in medical procedures with advantages of rapid action and minimal side effects.10% Lidocaine spray is a form of local anesthetic method that use in obstetrics and gynecology procedures and has favorable efficacy in reducing pain. Nevertheless, there were limited studies of 10% Lidocaine spray during IUD insertion. In this study, we investigate pain during IUD insertion using lidocaine spray compared with placebo.

ELIGIBILITY:
Inclusion Criteria:

* Woman who required for Copper T IUD insertion
* Body mass index 18.5 - 30 kg/m2
* Communicable with Thai language
* New IUD user

Exclusion Criteria:

* Suspicion of pregnancy
* Puerperal sepsis/Immediate post-septic abortion
* Untreated abnormal uterine bleeding
* Uterine anomaly/abnormal pathology distorting the uterine cavity
* Current pelvic inflammatory disease
* Untreated cervicitis/vaginitis
* Wilson's disease
* Copper allergy
* known hypersensitivity to local anaesthetic
* Analgesic or anxiolytic use within the last 24 h before the procedure

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 124 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2019-12-17 (Actual); Study Completion 2019-12-17 (Actual)

PRIMARY OUTCOMES:
Efficacy of 10% Lidocaine spray in reducing pain during IUD insertion: visual analog scale | Immediately after the procedure
  Assessment of pain using visual analog scale 0-10, 0 = minimum and 10 = maximum scores

SECONDARY OUTCOMES:
Side effects of 10% Lidocaine spray | 20 minutes after the procedure
  Presence or absence of side effects

CONTACTS AND LOCATIONS:
Overall Officials: Nalinee Panichyawat, Principal Investigator — Department of Obstetrics and Gynecology, Faculty of Medicine Siriraj hospital
Locations (1):
- Nalinee Panichyawat, Ratchathewi, Bangkok, Thailand

REFERENCES:
- [Derived] Panichyawat N, Mongkornthong T, Wongwananuruk T, Sirimai K. 10% lidocaine spray for pain control during intrauterine device insertion: a randomised, double-blind, placebo-controlled trial. BMJ Sex Reprod Health. 2021 Jul;47(3):159-165. doi: 10.1136/bmjsrh-2020-200670. Epub 2020 Jun 26. PMID 32591417